CLINICAL TRIAL: NCT01489956
Title: Pilot Study to Determine the Immunogenicity of Immucothel® and Oral Tolerance Induction With Biosyn Native KLH in Healthy Subjects (ITN047AI)
Brief Title: A Study to Determine the Immunogenicity and Oral Tolerance to Keyhole Limpet Hemocyanin (KLH)
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Due to futility, identified after 5 subjects completed treatment in Part B
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Immune Tolerance Network (ITN) (Network)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DAIT ITN047AI
Record Dates: First submitted 2011-12-01; First posted 2011-12-12 (Estimated); Results first posted 2016-04-12 (Estimated); Last update posted 2016-04-12 (Estimated); Status verified 2016-03

CONDITIONS: Autoimmune Disorders
Keywords: Keyhole Limpet Hemocyanin (KLH); Immucothel; Native KLH; Healthy volunteers; Oral tolerance; Immunogenicity; Autoimmune diseases
MeSH Terms: conditions — Autoimmune Diseases | interventions — keyhole-limpet hemocyanin; montanide ISA 51

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Immucothel alone (Part A) (Experimental): 100 µg Immucothel subcutaneously (SQ) on Day 0 and Day 9.
  Interventions: Biological: Immucothel Alone (Part A)
- Immucothel+Montanide (Part A) (Experimental): If an immune response was not observed in at least nine out of the first 10 participants after receiving Immucothel alone, 10 additional healthy subjects would be recruited and immunized with Immucothel (SQ) plus Montanide (SQ) on Day 0 and Day 9.
  Interventions: Biological: Immucothel+Montanide (Part A)
- Immucothel alone or Immucothel+Montanide (Part B) (Experimental): Dependent on the results for Part A.
  Briefly: Ten new, healthy participants were to be fed 50 mg of native keyhole limpet hemocyanin (KLH), a protein extracted from a mollusk (a sea animal), on Days 0 through 4 and Days 10 through 14, for a total dose of 500 mg. The participants were then immunized using the strategy that produced an immune response in at least nine out of 10 participants in Part A (Immucothel alone or Immucothel plus Montanide) on Days 26 and 35.
  Interventions: Biological: Immucothel Alone or Immucothel+Montanide (Part B)

INTERVENTIONS:
Biological: Immucothel Alone (Part A) — 100 ug at day 0 (priming dose) and day 9(booster dose)
  Other Names: keyhole limpet hemocyanin (KLH); Low Molecular Weight (LMW) KLH
  Arms: Immucothel alone (Part A)
Biological: Immucothel+Montanide (Part A) — 100 ug SQ Immucothel plus Montanide at day 0 (priming dose) and day 9 (booster dose)
  Other Names: Immucothel® + Montanide ISA 51; LMW KLH +oil based adjuvant
  Arms: Immucothel+Montanide (Part A)
Biological: Immucothel Alone or Immucothel+Montanide (Part B) — 50 mg of native KLH on days 0-4 and 10-14 (total of 500 mg). Immunization on days 26 and 35.
  Other Names: Immucothel® or Immucothel® + Montanide ISA 51; LMW KLH or LMW KLH +oil based adjuvant
  Arms: Immucothel alone or Immucothel+Montanide (Part B)

SUMMARY:
The purpose of this study is to test the oral tolerance of Keyhole Limpet Hemocyanin (KLH) and to determine if Immucothel by itself is strong enough to trigger the immune response. If not, Immucothel will be tested in combination with an adjuvant to determine if an adequate immune response can be seen.

DETAILED DESCRIPTION:
One type of normal immune response is called "oral tolerance." This is when the immune system (the body's natural defense system against illness) turns off (e.g. does not respond) to foods or to other proteins that are eaten. Oral tolerance test is done by feeding people a protein and then vaccinating them with the same protein. Oral tolerance occurs if the vaccination does not cause an immune response.

In this study, oral tolerance of Keyhole Limpet Hemocyanin (KLH) will be tested. KLH is a large protein extracted from a mollusk (a sea animal). The 'native KLH' (which is a large version of this protein) formulation will be used for oral feeding. Immucothel (a smaller version of the KLH protein) will be used for vaccination (injection). Immucothel is an investigational vaccine currently used to treat bladder cancers outside of the US.

Since these particular KLH products have never been used in oral tolerance studies, the investigators want to make sure in this pilot study that they will work as expected in healthy participants before studying these two products in patients with auto-immune disorders.

This study will also determine if Immucothel by itself is strong enough to trigger the immune response. If not, Immucothel will be tested in combination with an adjuvant (a substance that can increase the immune response to a protein like KLH) to determine if an adequate immune response can be seen.

This study consists of two parts. Participants will participate for either 39 days (Part A) or 65 days (Part B). Regardless of the group assignment, a safety follow-up phone call will occur 6 months after the last immunization (189 day for Part A or 215 day for part B) to assess the late onset of adverse events.

Part A of the study will test the experimental vaccine Immucothel by itself or in combination with an adjuvant. Immucothel is a purified protein from a mollusk. Immucothel can be given as a sub-q injection (under the skin) alone or with an adjuvant (a small amount of mineral oil) to help to enhance the immune response. There maybe two groups in this part:

1. Ten evaluable (as defined by protocol) participants will be given Immucothel alone by injection on two occasions, If Immucothel alone creates an immune response in most of the participants then Part A will be completed.
2. If Immucothel alone does not create an immune response in most of the participants in Part A, then 10 new evaluable (as defined by protocol) participants will be asked to volunteer to test Immucothel in combination with the adjuvant Montanide (mineral oil). This will be given by injection on two occasions If there is an immune response in most of the participants to this combination of Immucothel and Montanide then Part A will be done.

Part B of the study will test the successful Immucothel regimen from Part A with oral KLH. Ten new evaluable (as defined by protocol) participants will be given the experimental oral KLH.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Ability to give informed consent and comply with study procedures.
* Participant able/willing to hold off receiving prophylactic immunizations (like influenza or pneumococcal vaccines) during the study period.

Exclusion Criteria:

* Use of corticosteroids within 2 weeks prior to screening visit.
* First degree relative (parent, sibling or child) with history of autoimmune disease.
* Presence of chronic medical illness including but not limited to chronic kidney-, liver-, cardio-vascular diseases, immunodeficiencies, anemia, B12 deficiency, malignancies, or chronic active infections.
* History of acute gastrointestinal illness within 2 weeks prior to oral KLH administration.
* For women of child bearing age, participant unwilling to defer pregnancy, has a positive urine pregnancy test or is currently pregnant or lactating.
* Use of an investigational drug within 3 months of the screening visit.
* History of acute febrile illness within 1 week of screening visit.
* History of allergy to shellfish, previous exposure to KLH/product containing KLH or known-sensitivity to KLH / components of KLH preparation.
* Participants receiving any immunizations within 1 month prior to screening visit.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2011-12; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lloyd Mayer, MD, Study Chair — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mount Sinai Medical Center, New York, New York, United States

REFERENCES:
- See also: National Institute of Allergy and Infectious DiseasesDivision of Allergy, Immunology, and Transplantation (DAIT) — http://www.niaid.nih.gov/about/organization/dait/pages/default.aspx
- See also: National Institute of Allergy and Infectious Diseases — http://www.niaid.nih.gov/Pages/default.aspx
- See also: Immune Tolerance Network (ITN) — http://www.immunetolerance.org/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: One site in the United States recruited 19 healthy adult male and female participants.
Pre-assignment Details: The accrual objective was 10 to 20 evaluable participants in Part A and 10 evaluable participants in Part B. The definition of an evaluable participant (measured/determined by lymphocyte proliferation assay) was provided in the protocol.
Groups:
- Immucothel Alone (Part A): Subjects received 100 µg Immucothel subcutaneously (SQ) on Day 0 and Day 9. If at least nine of the subjects demonstrated an immune response, Part A of the study would be complete.
- Immucothel + Montanide (Part A): If an immune response was not observed in at least nine of the subjects after receiving Immucothel alone, 10 additional healthy subjects would be recruited and immunized with Immucothel (SQ) plus Montanide (SQ) on Day 0 and Day 9. If at least nine of the subjects had an immune response after receiving Immucothel plus Montanide, Part A of the study would be completed.
- Immucothel Alone or Immucothel + Montanide (Part B): Ten new, healthy participants ingested 50 mg of native keyhole limpet hemocyanin (KLH) orally. KLH, a protein extracted from a mollusk (a sea animal), was ingested on Days 0 through 4 and Days 10 through 14, for a total dose of 500 mg. The participants were then immunized using the strategy that produced an immune response in at least nine out of 10 participants in Part A (Immucothel alone or Immucothel plus Montanide) on Days 26 and 35.
Period: Overall Study
Arm/Group | Immucothel Alone (Part A) | Immucothel + Montanide (Part A) | Immucothel Alone or Immucothel + Montanide (Part B)
Started | 13 (Ten of the 13 participants were considered evaluable.) | 0 (Nine of the 10 participants receiving Immucothel alone had a response, so Montanide was not used.) | 6 (These 6 subjects had Immucothel alone since Montanide was not needed for the 10 participants dosed.)
Completed | 12 | 0 | 5
Not Completed | 1 | 0 | 1
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Enrolled Sample
Groups:
- Total: Total of all reporting groups
Arm/Group | Immucothel Alone (Part A) | Immucothel Alone or Immucothel + Montanide (Part B) | Total
Number analyzed (Participants) | 13 | 6 | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 13 | 6 | 19
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 5 | 13
  Male | 5 | 1 | 6
Region of Enrollment [Number; unit: participants]
  United States | 13 | 6 | 19

OUTCOME MEASURES:

1. Primary Outcome: Participants With a Positive Immune Response to T Cell Stimulation Index (SI) as Measured by 3H-thymidine Incorporation After in Vitro KLH Stimulation of PBMC (Part A)
Description: T cell stimulation index (SI) as measured by 3H-thymidine incorporation after in vitro keyhole limpet hemocyanin (KLH) stimulation of peripheral blood mononuclear cells (PBMC). An SI ≥3 on day 16 will indicate the presence of immune response. The SI is the ratio of 3H-thymidine incorporation by T cells in the presence of KLH stimulation to 3H-thymidine incorporation by T cells in the absence of stimulation. Higher values correspond with lower tolerance to KLH.
Time Frame: Day 16
Population: Intent-to-treat
Measure: Number; unit: participants
Arm/Group | Immucothel Alone (Part A) | Immucothel + Montanide (Part A) | Immucothel Alone or Immucothel + Montanide (Part B)
Number analyzed (Participants) | 10 | 0 | 0
participants | 9 |  |

2. Primary Outcome: Participants Demonstrating Tolerance to KLH Using T Cell Stimulation Index (SI) as Measured by 3H-thymidine Incorporation After in Vitro KLH Stimulation of PBMC (Part B)
Description: T cell stimulation index (SI) as measured by 3H-thymidine incorporation after in vitro keyhole limpet hemocyanin (KLH) stimulation of peripheral blood mononuclear cells (PBMC). An SI <3 on Day 32 indicated tolerance to KLH. The SI is the ratio of 3H-thymidine incorporation by T cells in the presence of KLH stimulation to 3H-thymidine incorporation by T cells in the absence of stimulation. Higher values correspond with lower tolerance to KLH.
Time Frame: Day 32
Population: Intent-to-treat
Measure: Number; unit: participants
Arm/Group | Immucothel Alone (Part A) | Immucothel + Montanide (Part A) | Immucothel Alone or Immucothel + Montanide (Part B)
Number analyzed (Participants) | 0 | 0 | 5
participants |  |  | 1

3. Primary Outcome: T Cell Stimulation Index (SI) as Measured by 3H-thymidine Incorporation After in Vitro KLH Stimulation of PBMC (Part A)
Description: No data available for analyses
Time Frame: Day 9
Population: Data were not collected and therefore no analyses could be performed.
Arm/Group | Immucothel Alone (Part A) | Immucothel + Montanide (Part A) | Immucothel Alone or Immucothel + Montanide (Part B)
Number analyzed (Participants) | 0 | 0 | 0

4. Primary Outcome: T Cell Stimulation Index (SI) as Measured by 3H-thymidine Incorporation After in Vitro KLH Stimulation of PBMC (Part A)
Description: No data available for analyses.
Time Frame: Day 16
Population: Data were not collected and therefore no analyses could be performed.
Arm/Group | Immucothel Alone (Part A) | Immucothel + Montanide (Part A) | Immucothel Alone or Immucothel + Montanide (Part B)
Number analyzed (Participants) | 0 | 0 | 0

5. Secondary Outcome: Cytokine Secretion Profile of T Cells Stimulated by KLH (Part A)
Description: No data available for analyses.
Time Frame: Days 0, 9, 16
Population: Data were not collected and therefore no analyses could be performed.
Arm/Group | Immucothel Alone (Part A) | Immucothel + Montanide (Part A) | Immucothel Alone or Immucothel + Montanide (Part B)
Number analyzed (Participants) | 0 | 0 | 0

6. Secondary Outcome: T Cell Stimulation Index Measured by Carboxyfluorescein Diacetate Succinimidyl Ester (CFSE) Staining After KLH Stimulation (Part A)
Description: No data available for analyses.
Time Frame: Days 0, 9, 16
Population: Data were not collected and therefore no analyses could be performed.
Arm/Group | Immucothel Alone (Part A) | Immucothel + Montanide (Part A) | Immucothel Alone or Immucothel + Montanide (Part B)
Number analyzed (Participants) | 0 | 0 | 0

7. Secondary Outcome: Suppression (or Non-activation) of Cytokine Secretion Profile of T Cells Stimulated by KLH Following Oral Feeding (Part B)
Description: No data available for analyses.
Time Frame: Day 42
Population: Data were not collected and therefore no analyses could be performed.
Arm/Group | Immucothel Alone (Part A) | Immucothel + Montanide (Part A) | Immucothel Alone or Immucothel + Montanide (Part B)
Number analyzed (Participants) | 0 | 0 | 0

8. Secondary Outcome: Suppression (or Non-activation) of T Cell Stimulation Index Measured by CFSE Staining After KLH Stimulation (Part B)
Description: No data available for analyses.
Time Frame: Day 42
Population: Data were not collected and therefore no analyses could be performed.
Arm/Group | Immucothel Alone (Part A) | Immucothel + Montanide (Part A) | Immucothel Alone or Immucothel + Montanide (Part B)
Number analyzed (Participants) | 0 | 0 | 0

9. Secondary Outcome: Other Mechanistic Assessments on Archived Serum Samples Like Anti-KLH Antibodies and Secreted Cytokines (Part B)
Description: No data available for analyses.
Time Frame: 6 months
Population: Data were not collected and therefore no analyses could be performed.
Arm/Group | Immucothel Alone (Part A) | Immucothel + Montanide (Part A) | Immucothel Alone or Immucothel + Montanide (Part B)
Number analyzed (Participants) | 0 | 0 | 0

10. Secondary Outcome: Compare the Level of KLH-specific Antibodies in the Serum (Samples From Various Time Points) Between Parts A and B
Description: No data available for analyses.
Time Frame: 6 months
Population: Data were not collected and therefore no analyses could be performed.
Arm/Group | Immucothel Alone (Part A) | Immucothel + Montanide (Part A) | Immucothel Alone or Immucothel + Montanide (Part B)
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Enrollment through last study visit (up to 6 months after last immunization)
Description: Adverse events reported for all enrolled subjects
Arm/Group | Immucothel Alone (Part A) | Immucothel + Montanide (Part A) | Immucothel Alone or Immucothel + Montanide (Part B)
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/0 | 0/6
Other Adverse Events (participants affected / at risk) | 4/13 | 0/0 | 4/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Immucothel Alone (Part A) (N=13) | Immucothel + Montanide (Part A) (N=0) | Immucothel Alone or Immucothel + Montanide (Part B) (N=6)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Injection site reaction (General disorders) | 0 (0) | 0 (0) | 1 (1)
Gingival infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Basophil count increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Basophil percentage increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Eosinophil percentage increased (Investigations) | 0 (0) | 0 (0) | 1 (2)
Haematocrit decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Haematocrit increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Haemoglobin decreased (Investigations) | 2 (2) | 0 (0) | 0 (0)
Haemoglobin increased (Investigations) | 0 (0) | 0 (0) | 2 (3)
Mean cell haemoglobin decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Red blood cell count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 1 (1) | 0 (0) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Breast reconstruction (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Data from 4 of the 5 evaluable subjects in Part B was negative for tolerance to KLH as defined by a stimulation index <3 on day 42 after booster immunization. The study was terminated. Data were not collected and no analyses were performed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No